CLINICAL TRIAL: NCT03700047
Title: A Randomized, Evaluator-Blinded, Parallel, Comparator-Controlled Study to Evaluate the Safety and Effectiveness of GAL1704 for Cheek Augmentation and Correction of Midface Contour Deficiencies
Brief Title: GAL1704 for Cheek Augmentation and Correction of Midface Contour Deficiencies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43USV1704
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Results first posted 2022-05-31 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-05

CONDITIONS: Cheek Augmentation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- GAL1704 (needle) (Experimental): Subjects randomized (2:1) to GAL1704 or Control for cheek augmentation and the correction of midface contour deficiencies.
  Interventions: Device: GAL1704
- GAL1704 (cannula/needle) (Experimental): GAL1704 treatment using a split face design - one cheek treated using cannula and the other cheek treated using needle.
  Interventions: Device: GAL1704
- Juvederm Voluma (Active Comparator): Subjects randomized to control.
  Interventions: Device: Juvederm Voluma

INTERVENTIONS:
Device: GAL1704 — new dermal filler
  Arms: GAL1704 (cannula/needle); GAL1704 (needle)
Device: Juvederm Voluma — hyaluronic acid
  Arms: Juvederm Voluma

SUMMARY:
An interventional study to evaluate the safety and effectiveness of GAL1704 for cheek augmentation and the correction of midface volume deficiencies by demonstrating non-inferiority in change from baseline, relative to an active comparator.

ELIGIBILITY:
Inclusion Criteria:

- Subjects assessed at baseline by the Blinded Evaluator as Grade 2, 3, or 4 on the MMVS on each side of the midface.

Exclusion Criteria:

- Previous use of any HA based or collagen based biodegradable tissue augmentation therapy within 12 months prior to the baseline visit

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2020-05-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Galderma Study site, Los Angeles, California
  - Galderma Study Site, Sacramento, California
  - Galderma Study Site, Solana Beach, California
  - Galderma Study Site, Miami, Florida
  - Galderma Study Site, West Palm Beach, Florida
  - Galderma Study Site, New Orleans, Louisiana
  - Galderma Study Site, Baltimore, Maryland
  - Galderma Study Site, Chestnut Hill, Massachusetts
  - Galderma Study Site, Mount Kisco, New York
  - Galderma Study Site, New York, New York
  - Galderma study site, Charleston, South Carolina
  - Galderma study site, Bellaire, Texas
  - Galderma Study site, Dallas, Texas
  - Galderma Study Site, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GAL1704 (Needle) | GAL1704 (Cannula/Needle) | Juvederm Voluma
Started | 142 | 60 | 68
Completed | 126 | 50 | 58
Not Completed | 16 | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- GAL1704 (Cannula): GAL1704 treatment using a split face design - one cheek treated using cannula and the other cheek treated using needle
- Total: Total of all reporting groups
Arm/Group | GAL1704 (Needle) | GAL1704 (Cannula) | Juvederm Voluma | Total
Number analyzed (Participants) | 142 | 60 | 68 | 270
Age, Continuous [Mean (Full Range); unit: years] | 52.7 [24 to 79] | 52.1 [28 to 73] | 54.7 [24 to 80] | 52.7 [24 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 55 | 58 | 242
  Male | 13 | 5 | 10 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 2 | 3 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 8 | 13 | 7 | 28
  White | 125 | 44 | 57 | 226
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 142 | 60 | 68 | 270
Fitzpatrick Skin Type (FST) [Count of Participants; unit: Participants] — FST is a standardized skin classification system with 6 skin phototypes, where FST I represents the lightest skin color and FST VI represents the darkest skin color.
  Participants
    FST I | 4 | 1 | 1 | 6
    FST II | 40 | 9 | 23 | 72
    FST III | 65 | 27 | 28 | 120
    FST IV | 17 | 8 | 9 | 34
    FST V | 8 | 3 | 3 | 14
    FST VI | 8 | 12 | 4 | 24

OUTCOME MEASURES:

1. Primary Outcome: Assess Efficacy of Study Treatment Using Medicis Midface Volume Score (MMVS)
Description: Change in midface fullness from Baseline to 12 weeks using the Medicis Midface Volume Score (MMVS), where a decreasing score correlates with increasing midface fullness, namely a score of 1 being the most full and a score of 4 being the least full.
Time Frame: 12 weeks
Population: Per protocol population
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | GAL1704 (Needle) | GAL1704 (Cannula/Needle) | Juvederm Voluma
Number analyzed (Participants) | 142 | 58 | 68
score on a scale | -1.4 [-1.51 to -1.35] | -0.1 [-0.16 to 0.05] | -1.3 [-1.44 to -1.20]

ADVERSE EVENTS:
Time Frame: 1 year, 2 months
Arm/Group | GAL1704 (Needle) | GAL1704 (Cannula/Needle) | Juvederm Voluma
All-Cause Mortality (participants affected / at risk) | 0/142 | 0/60 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/141 | 1/60 | 2/68
Other Adverse Events (participants affected / at risk) | 6/141 | 0/60 | 13/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GAL1704 (Needle) (N=141) | GAL1704 (Cannula/Needle) (N=60) | Juvederm Voluma (N=68)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GAL1704 (Needle) (N=141) | GAL1704 (Cannula/Needle) (N=60) | Juvederm Voluma (N=68)
Implant site pain (General disorders) | 6 (16) | 0 (0) | 13 (49)
Implant site oedema (General disorders) | 3 (6) | 0 (0) | 7 (19)
Implant site erythema (General disorders) | 2 (6) | 0 (0) | 6 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs agree not to present or publish any data or reports collected individually or by subgroup of sites prior to full, initial publication based on all data obtained from all sites.

DOCUMENTS (2):
  • Study Protocol (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT03700047/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT03700047/SAP_001.pdf